CLINICAL TRIAL: NCT04380363
Title: Safety and Usability Assessment of the Honda Walking Assist Device (HWA) for Personal Use in Home and Community Environments
Brief Title: Safety and Usability of the Honda Walking Assist Device (HWA) in the Home Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Honda Research and Development Americas (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00211619
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Stroke; Gait; Honda Walk Assist
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects randomized into device or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Honda Walk Assist (HWA) Group (Experimental): Participants utilize HWA device at home for 2 months according to prescribed settings.
  Interventions: Device: Honda Walk Assist (HWA) device
- Control Group (Active Comparator): Participants complete prescribed exercise program at the Shirley Ryan AbilityLab gym for 2 months.
  Interventions: Other: SRALab fitness center membership

INTERVENTIONS:
Device: Honda Walk Assist (HWA) device — Use of HWA for 2 months in the home setting
  Arms: Honda Walk Assist (HWA) Group
Other: SRALab fitness center membership — Membership to Shirley Ryan AbilityLab fitness center for 2 months
  Arms: Control Group

SUMMARY:
The purpose of this study is to verify the safety and validate the usability of the Honda Walk Assist (HWA) device in the home setting versus an exercise program without the device in a gym setting for individuals diagnosed with stroke. The investigators hypothesize that the HWA exoskeleton is a safe and effective device for use by individuals diagnosed with stroke in the home environment.

DETAILED DESCRIPTION:
The purpose of this randomized control trial is to determine the safety and usability of the Honda Walk Assist (HWA) device in the home environment versus a gym membership. Secondarily, the study will investigate effects of the HWA exoskeleton in the home environment versus a gym membership on gait function and overall home training activity. Participants who are greater than 1 year post stroke and between the ages of 18-80 will be included.

The HWA device is a lightweight, robotic exoskeleton designed to support people with gait deficits. The device is worn around the user's torso, waist and thighs, and assists with hip flexion and extension. The device weighs about 6lbs and has two motors that run on a single rechargeable battery. The device is equipped with angle and current sensors to monitor hip joint angle and torque output respectively. The adjustable assist torque (6Nm max.) is transmitted to the user's thighs via thigh frames. A trained healthcare professional can initially configure assist settings through software that runs on a mobile device. This trained professional can also make device adjustments to ensure a proper fit for the user and train the user for personal use of the HWA. After initial settings are established, users can don, doff and operate the device independently or with the help of an assistant.

Participant with stroke greater than 1 year ago will be recruited from outpatient clinics, day rehabilitation sites, and the hospital's research registry. Following a screening session to determine subject eligibility, subjects will be randomized to either the HWA or gym membership groups.

Baseline outcome measures will be collected and subjects will wear an ActiGraph activity monitor for 1-2 weeks. Subjects will then complete 1-3 sessions with a research physical therapist to acclimate and individualize the HWA device's settings or will be introduced to the Shirley Ryan AbilityLab gym and prescribed an individualized exercise program. During the 2 month intervention, subjects will either utilize the HWA device at home according to the prescribed settings or complete the prescribed exercise program at the Shirley Ryan AbilityLab fitness center. Weekly phone calls from the physical therapists will check in on both groups to determine whether participants are following their exercise programs and to answer any questions or concerns. At the conclusion of the 2 month intervention, participants will wear an ActiGraph monitor for 1-2 weeks and outcome measures will again be collected over 2 testing visits.

All testing and acclimation sessions will be performed under the supervision of a licensed physical therapist. Adverse events will be recorded.

The investigators anticipate this study will help determine the feasibility of using the Honda Walk Assist device in the home setting in individuals greater than a year post stroke. The investigators do not foresee any potential pitfalls.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year post stroke
* initial gate speed of > 0.2 m/s and < 0.8 m/s
* adequate cognitive function (MMSE score >17)
* subject is willing to be randomized to the control group or the treatment group
* ability to sit unsupported for 30 seconds
* ability to walk at least 10m without physical assist
* ability to follow a 3-step command
* physician approval for patient participation
* living in the community post-stroke with the ability to travel to the intervention site to participate in the outpatient program and able to perform the home exercise program in a residential facility

Exclusion Criteria:

* participants who cannot move their limbs through the physical limits of the device (range of motion)
* less than 90 days post major orthopedic surgery (i.e. hip, knee, and/or ankle joint replacement)
* less than 6 months post CABG or cardiac valve procedure
* serious medical conditions including myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living, severe hypertension, severe weight bearing pain, life expectancy less than one year
* preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia
* history of major head trauma, lower extremity amputation, non-healing ulcers of a lower extremity, renal dialysis or end stage liver disease, legal blindness or severe visual impairment, a history of significant psychiatric illness
* pacemakers, metal implants in the head region
* subject is pregnant, nursing or planning a pregnancy
* expressive aphasia
* participating in another clinical trial that, according to the Principal Investigator, is likely to affect study outcome or confound results
* inability to perform 5 times per week for the home rehabilitation program
* individuals who need to use a walker with the device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HWA Device Log | 2 months of at-home training
  The HWA device is equipped with sensors that can detect hip joint angle movement. This joint angle data can be downloaded to an external computer. In the HWA group, HWA log data could provide an objective measure of participant activity when the HWA device is activated. HWA will be solely responsible for managing log data and will provide information of device use and misuse among therapists and study participants. This will also help determine device malfunctions.
Honda Training Experience Survey | 2 months of at-home training
  Each participant in the HWA group will be given a tablet to obtain subjective feedback about the HWA device and home training experience. These tablets will contain pre-loaded questions for subjects to answer on a daily basis to obtain information about device usability in the home setting.
10 Meter Walk Test (10MWT) | Baseline; Post-testing (after 2 month intervention)
  The 10MWT assesses walking speed in meters per second over a short duration of 10 meters (33 ft). In the 10MWT, subjects are directed to walk at their self-selected and maximum safe speed with the effects of acceleration and deceleration minimized by adding 1 meter at the beginning and at the end of the course to isolate the subject's steady state speed. Any assistive device and orthotic are kept consistent and documented. Gait speed at both the "self-selected walking speed" or "fastest walking speed" are recorded. The 10MWT has been validated for the stroke population and is accepted as a responsive, functional measurement of the patient's ability to ambulate over short distances such as those typical to a household setting.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Baseline; Post-testing (after 2 month intervention)
  The 6MWT measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The distance is measured with a measuring wheel. The instructions are "Walk covering as much ground as you can in 6 min. You can stop to sit or stand if needed, but time will keep running." The change in the distance walked in the 6-minute walk can be used to evaluate the efficacy of an exercise-training program or to trace the natural history of change in exercise capacity over time. The 6MWT is measured in meters. For the HWA intervention group, this will be tested both with and without use of the HWA device.
Gait Analysis | Baseline; Post-testing (after 2 month intervention)
  A quantitative means of assessing gait function in adults post-stroke based on spatiotemporal parameters of gait. The GAITRite® system is an electronic walkway with integrated sensors and is considered a reliable and valid means of assessing gait changes post-stroke. For the HWA intervention group, this will be tested both with and without use of the HWA device.
Functional Gait Assessment (FGA) | Baseline; Post-testing (after 2 month intervention)
  The FGA is a 10-item test for assessing postural stability during various walking tasks. It includes 7 of the 8 items from the original Dynamic Gait Index, and 3 new items, including "gait with narrow base of support", "ambulating backwards", and "gait with eyes closed". The FGA demonstrates excellent concurrent validity with the Berg Balance Scale for individuals with stroke. The maximum score is 30 points; minimal detectable change for chronic stroke is 4.2 points.
Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA) | Baseline; Post-testing (after 2 month intervention)
  The purpose of the FMA is to evaluate and measure recovery in post-stroke hemiplegic patients. There are five domains assessed on a 3-point ordinal scale from 0-2. "0" is equal to "cannot perform", "1" is equal to "performs partially", and "2" is equal to "performs fully". The domain for lower extremity motor function will be used. It has been found to be reliable and valid in assessing individuals with stroke with a minimal clinically important difference of 10 points for the lower extremity motor scores.
Manual Muscle Testing (MMT) | Baseline; Post-testing (after 2 month intervention)
  The purpose of this test is to evaluate the strength of the legs by having the subject hold the legs in a position while the researcher applies manual resistance.
Modified Ashworth Test (MAS) | Baseline; Post-testing (after 2 month intervention)
  The purpose of this test is to evaluate the amount of spasticity in the legs.
Passive Range of Motion (PROM) | Baseline; Post-testing (after 2 month intervention)
  The purpose of this test is to evaluate a subject's passive range of motion in the joints of the hips, knees and ankles.
Activites-Specific and Balance Confidence Scale (ABC) | Baseline; Post-testing (after 2 month intervention)
  The ABC is a 16-item self-report questionnaire that measures confidence in performing various ambulatory activities without falling. Items are rated on a scale ranging from 0-100, with zero representing no confidence and 100 representing complete confidence. It has good to excellent reliability and adequate construct validity, correlating with the BBS and 10MWT.
Stroke Specific Quality of Life (SSQoL) | Baseline; post-testing (after 2 month intervention)
  The SSQoL is a self-report questionnaire that is accepted as a reliable and valid way to assess health-related quality of life specific to stroke survivors. Subjects respond to 49 questions in 12 domains: mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality. Each individual domain consists of 3 to 10 items that are averaged to generate an overall score, each item is rated on a 5- point Likert scale, with a minimum value of 1 (meaning the worst outcome) and a maximum value of 5 (meaning the best outcome). Domains scores (non-weighted average of item scores) and a summary score (non-weighted average of all 12 domain scores) are computed. Summary scores range from 49-245, with higher scores indicating better functioning.
Physical Therapist Interview | Post-testing (after 2 month intervention)
  During the final post-test session at SRAlab, therapists will ask participants various questions about their experience throughout the study. This could be through a verbal discussion or through a written questionnaire. The purpose of this interview is to collect subjective feedback from therapists and study participants regarding overall impressions of device use.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No